CLINICAL TRIAL: NCT05163288
Title: Effects of N-Acetyl-L-Leucine on Niemann-Pick Disease Type C (NPC): A Phase III, Randomized, Placebo-controlled, Double-blind, Crossover Study
Brief Title: A Pivotal Study of N-Acetyl-L-Leucine on Niemann-Pick Disease Type C
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IntraBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IB1001-301
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Niemann-Pick Disease, Type C
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — acetylleucine; IB1001

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, crossover, multi-center, study with 1:1 randomization of IB1001 plus SOC for 12-weeks versus placebo plus SOC for 12-weeks, followed by open-label extension study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetyl-L-leucine (IB1001) (Experimental): Oral administration (granule in a sachet for suspension in water, orange juice, or almond milk). Patients ≥13 years old will receive a total daily dose of 4 g/day (administered as 3 doses per day); patients <13 will receive weight-tiered doses.
  Interventions: Drug: N-Acetyl-L-Leucine
- Placebo comparator (Placebo Comparator): Oral administration (granule in a sachet for suspension in water, orange juice, or almond milk). Patients ≥13 years old will receive a total daily dose of 4 g/day (administered as 3 doses per day); patients <13 will receive weight-tiered doses.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: N-Acetyl-L-Leucine — N-Acetyl-L-Leucine is a modified amino-acid ester that is orally administered (granules for suspension in a sachet)
  Other Names: IB1001
  Arms: N-acetyl-L-leucine (IB1001)
Other: Placebo — Matching Placebo Sachet
  Arms: Placebo comparator

SUMMARY:
A pivotal, randomized, double-blind, placebo controlled, multi-center therapeutic study for patients age 4 and older with a confirmed diagnosis of Niemann Pick disease type C (NPC). The objective of this study is to evaluate the safety, tolerability and efficacy of N-acetyl-L-leucine (IB1001) compared to standard of care.

Following this randomized, double-blind, placebo-controlled "Parent Study", an extension phase is conducted for (1) patients who completed the "Parent Study" and (2) patients who are enrolled directly into the Extension Phase. Currently, the Extension Phase provides patients with 3 years of open-label treatment.

DETAILED DESCRIPTION:
This is a multinational, randomized, placebo-controlled, double-blinded, cross-over Phase III study that will assess the safety and efficacy of N-Acetyl-L-Leucine (IB1001) versus Placebo for the treatment of Niemann-Pick type C disease (NPC).

Patients will be assessed during three study periods: a baseline period (approximately 2-weeks), after which they will be randomized (1:1) to receive treatment with IB1001 or Placebo for approximately 12-weeks during the first intervention period ("Period I"). Following Period I, patients will crossover to receive the opposite treatment (IB1001 or Placebo) for approximately 12-weeks during a second intervention period ("Period II).

Patients will be assessed twice during each study period. Patients who have participated in the study may be offered the opportunity to roll over into an Extension Phase, which is planned to allow patients to have further access to IB1001.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed by the patient and/or their legal representative/ parent/ impartial witness
2. Male or female aged ≥4 years with a confirmed genetic diagnosis of NPC at the time of signing informed consent.
3. Females of childbearing potential, defined as a premenopausal female capable of becoming pregnant, will be included if they are either sexually inactive (sexually abstinent for 14 days prior to the first dose and confirm to continue through 28 days after the last dose) or using one of the following highly effective contraceptives (i.e. results in <1% failure rate when used consistently and correctly) 14 days prior to the first dose continuing through 28 days after the last dose:

   1. intrauterine device (IUD);
   2. surgical sterilization of the partner (vasectomy for 6 months minimum);
   3. combined (estrogen or progestogen containing) hormonal contraception associated with the inhibition of ovulation (either oral, intravaginal, or transdermal);
   4. progestogen only hormonal contraception associated with the inhibition of ovulation (either oral, injectable, or implantable);
   5. intrauterine hormone releasing system (IUS);
   6. bilateral tubal occlusion.
4. Females of non-childbearing potential who have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

   1. hysteroscopic sterilization;
   2. bilateral tubal ligation or bilateral salpingectomy;
   3. hysterectomy;
   4. bilateral oophorectomy; OR be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status. FSH analysis for postmenopausal women will be done at screening. FSH levels should be in the postmenopausal range as determined by the central laboratory.
5. Non-vasectomized male patient agrees to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study medication and the female partner agrees to comply with inclusion criteria 3 or 4.

   For a vasectomized male who has had his vasectomy 6 months or more prior to study start, it is required that they use a condom during sexual intercourse. A male who has been vasectomized less than 6 months prior to study start must follow the same restrictions as a non-vasectomized male.
6. If male, patient agrees not to donate sperm from the first dose until 90 days after their last dose.
7. Patients must fall within:

   a) A SARA score of 7 ≤ X ≤ 34 points (out of 40) AND b) Either: i. Within the 2-7 range (0-8 range) of the Gait subtest of the SARA scale OR ii. Be able to perform the 9-Hole Peg Test with Dominant Hand (9HPT-D) (SCAFI subtest) in 20 ≤ X ≤150 seconds.
8. Weight ≥15 kg at screening.
9. Patients are willing to disclose their existing medications/therapies for (the symptoms) of NPC including those on the prohibited medication list. Non-prohibited medications/therapies (authorized medicines for NPC [e.g. miglustat], speech therapy, and physiotherapy) are permitted provided:

   1. The Investigator does not believe the medication/therapy will interfere with the study protocol/results
   2. Patients have been on a stable dose/duration and type of therapy for at least 42 days before Visit 1 (Baseline 1)
   3. Patients are willing to maintain a stable dose/do not change their therapy throughout the duration of the study.
10. An understanding of the implications of study participation, provided in the written patient information and informed consent by patients or their legal representative/parent, and demonstrates a willingness to comply with instructions and attend required study visits (for children this criterion will also be assessed in parents or appointed guardians).

Exclusion Criteria:

1. Patients who are unable to consistently Patients who have any known hypersensitivity or history of hypersensitivity to:

   1. Acetyl-Leucine (DL-, L-, D-) or derivatives.
   2. Excipients the IB1001 sachet (namely isomalt, hypromellose, and strawberry flavour).
   3. Excipients the placebo sachet (namely isomalt, hypromellose, strawberry flavour, citric acid, microcrystalline cellulose, lactose, denatonium benzoate).
2. Simultaneous participation in another clinical study or participation in any clinical study involving administration of an investigational medicinal product (IMP; 'study drug') for at least 42 days prior to Visit 1. At the discretion of the investigator, Medical Monitor, and Sponsor, the washout period for specific IMPs may be longer based on the pharmacological activity and pharmacokinetics of the drug.
3. Patients with a physical, cognitive, or psychiatric condition which, at the investigator's discretion and in consultation with the Medical Monitor and Sponsor (as applicable), may put the patient at risk, may confound the study results, or may interfere with the patient's participation in the clinical study, i.e. reliably perform study assessments.
4. Known or persistent use, misuse, or dependency of medication, drugs, or alcohol.
5. Current or planned pregnancy or women who are breastfeeding.
6. Patients with severe vision or hearing impairment (that is not corrected by glasses or hearing aids) that, at the investigator's discretion, interferes with their ability to perform study assessments.
7. Patients who have been diagnosed with arthritis or other musculoskeletal disorders affecting joints, muscles, ligaments, and/or nerves that by themselves affects patient's mobility and, at the investigator's discretion, interferes with their ability to perform study assessments.
8. Patients unwilling and/or not able to undergo a 42 day period from any of the following prohibited medication prior to Visit 1 (Baseline 1) and remain without prohibited medication through Visit 6.

   1. N-Acetyl-DL-Leucine (e.g. Tanganil®);
   2. N-Acetyl-L-Leucine (prohibited if not provided as IMP in the IB1001-301 trial);
   3. Sulfasalazine;
   4. Rosuvastatin.

      -

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (all jurisdictions except US) | End of Period I (week 12) vs. End of Period 2 (week 24)
Modified Scale for the Assessment and Rating of Ataxia (US only) | End of Period I (week 12) vs. End of Period 2 (week 24)

SECONDARY OUTCOMES:
Spinocerebellar Ataxia Functional Index (SCAFI) | End of Period I (week 12) vs. End of Period 2 (week 24)
Modified Disability Rating Scale | End of Period I (week 12) vs. End of Period 2 (week 24)
Physician's / Caregiver's / Patient's Clinical Global Impressions (CGI) | End of Period I (week 12) vs. End of Period 2 (week 24)
EuroQuol- 5 Dimension (EQ-5D) Quality of Life Scale | End of Period I (week 12) vs. End of Period 2 (week 24)
Scale for the Assessment and Rating of Ataxia (US only) | End of Period I (week 12) vs. End of Period 2 (week 24)

OTHER OUTCOMES:
Niemann-Pick disease type C Clinical Severity Scale (NPC-CSS) | End of Period I (week 12) vs. End of Period 2 (week 24)
5-Domain Niemann-Pick disease type C Clinical Severity Scale (NPC-CSS) | End of Period I (week 12) vs. End of Period 2 (week 24)
Investigator's / Caregiver's / Patient's Clinical Global Impressions (CGI) | End of Period I (week 12) vs. End of Period 2 (week 24)
Modified Scale for the Assessment and Rating of Ataxia (all jurisdictions except US) | End of Period I (week 12) vs. End of Period 2 (week 24)

CONTACTS AND LOCATIONS:
Locations (14):
- Mayo Clinic, Rochester, Minnesota, United States
- The Royal Melbourne Hospital, Parkville, Victoria, Australia
- First Faculty of Medicine, Charles University Hospital Prague, Prague, Czechia
- Germany (5):
  - University of Giessen, Giessen
  - University of Hamburg, Hamburg
  - SphinCS - Institute of Clinical Science in Lysosomal Storage Disorders, Höchheim
  - Ludwig Maximilian University of Munich, München
  - University Hospital Münster, Münster
- Amsterdam UMC, Amsterdam, Netherlands
- Comenius University in Bratislva, Bratislava, Slovakia
- University Hospital Bern Inselspital, Bern, Switzerland
- United Kingdom (3):
  - Great Ormond Street Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No
The results of the study will be published within a reasonable timeframe of completion. Pseudonymised individual patient data may be available in these findings.

REFERENCES:
- [Background] Bremova-Ertl T, Claassen J, Foltan T, Gascon-Bayarri J, Gissen P, Hahn A, Hassan A, Hennig A, Jones SA, Kolnikova M, Martakis K, Raethjen J, Ramaswami U, Sharma R, Schneider SA. Efficacy and safety of N-acetyl-L-leucine in Niemann-Pick disease type C. J Neurol. 2022 Mar;269(3):1651-1662. doi: 10.1007/s00415-021-10717-0. Epub 2021 Aug 13. PMID 34387740
- [Background] Kaya E, Smith DA, Smith C, Morris L, Bremova-Ertl T, Cortina-Borja M, Fineran P, Morten KJ, Poulton J, Boland B, Spencer J, Strupp M, Platt FM. Acetyl-leucine slows disease progression in lysosomal storage disorders. Brain Commun. 2020 Dec 20;3(1):fcaa148. doi: 10.1093/braincomms/fcaa148. eCollection 2021. PMID 33738443
- [Background] Cortina-Borja M, Te Vruchte D, Mengel E, Amraoui Y, Imrie J, Jones SA, I Dali C, Fineran P, Kirkegaard T, Runz H, Lachmann R, Bremova-Ertl T, Strupp M, Platt FM. Annual severity increment score as a tool for stratifying patients with Niemann-Pick disease type C and for recruitment to clinical trials. Orphanet J Rare Dis. 2018 Aug 16;13(1):143. doi: 10.1186/s13023-018-0880-9. PMID 30115089
- [Derived] Patterson MC, Ramaswami U, Donald A, Foltan T, Gautschi M, Gissen P, Hahn A, Jones SA, Kay R, Kolnikova M, Park J, Reichmannova S, Walterfang M, Wibawa P, Rohrbach M, Martakis K, Bremova-Ertl T. Disease-Modifying, Neuroprotective Effect of N-Acetyl-l-Leucine in Adult and Pediatric Patients With Niemann-Pick Disease Type C. Neurology. 2025 Jul;105(1):e213589. doi: 10.1212/WNL.0000000000213589. Epub 2025 Jun 13. PMID 40513057
- [Derived] Bremova-Ertl T, Ramaswami U, Brands M, Foltan T, Gautschi M, Gissen P, Gowing F, Hahn A, Jones S, Kay R, Kolnikova M, Arash-Kaps L, Marquardt T, Mengel E, Park JH, Reichmannova S, Schneider SA, Sivananthan S, Walterfang M, Wibawa P, Strupp M, Martakis K. Trial of N-Acetyl-l-Leucine in Niemann-Pick Disease Type C. N Engl J Med. 2024 Feb 1;390(5):421-431. doi: 10.1056/NEJMoa2310151. PMID 38294974